CLINICAL TRIAL: NCT06686290
Title: Effects of Post-Isometric Relaxation Versus Static Stretching on Pain, Range of Motion, Disability and Muscle Length in Patients With Levator Scapulae Syndrome.
Brief Title: Effects of Post-Isometric Relaxation Versus Static Stretching in Patients With Levator Scapulae Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0117
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Levator Scapulae Syndrome
Keywords: Disability; Range of Motion; Muscle Length; Pain
MeSH Terms: conditions — Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Group A will be treated with Postisometric relaxation technique and Group B will be treated with Static stretching technique. Postisometric relaxation will be performed with the frequency of 5 times, such that it includes (30 isometric contraction of the muscle to be stretched for 10 seconds, followed by rest period of 5 seconds and then a stretch of 10 seconds hold. Stretching exercise will be performed with 30 second hold and with 5 repetitions. All Exercises will be performed 3 times per week for total of 4 weeks.
Who Masked: Outcomes Assessor
Masking Description: Assessor Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Isometric Relaxation Technique (Experimental): Postisometric relaxation will be performed with the frequency of 5 times, such that it includes 30 isometric contraction of the muscle to be stretched for 10 seconds, followed by rest period of 5 seconds and then a stretch of 10 seconds hold.
  Interventions: Other: Post-Isometric Relaxation Technique
- Static Stretching (Experimental): Stretching exercise will be performed with 30 second hold and with 5 repetitions. All Exercises will be performed 3 times per week for total of 4 weeks.
  Interventions: Other: Static Stretching

INTERVENTIONS:
Other: Post-Isometric Relaxation Technique — Post isometric relaxation will be performed with the frequency of 5 times, such that it includes 30 isometric contraction of the muscle to be stretched for 10 seconds, followed by rest period of 5 seconds and then a stretch of 10 seconds hold.
  Arms: Post Isometric Relaxation Technique
Other: Static Stretching — Static Stretching
  Arms: Static Stretching

SUMMARY:
Group A will be treated with Postisometric relaxation technique and Group B will be treated with Static stretching technique. Postisometric relaxation will be performed with the frequency of 5 times, such that it includes (30 isometric contraction of the muscle to be stretched for 10 seconds, followed by rest period of 5 seconds and then a stretch of 10 seconds hold. Stretching exercise will be performed with 30 second hold and with 5 repetitions. All Exercises will be performed 3 times per week for total of 4 weeks. Outcome measures will be conducted through pain, range of motion, disability and muscle length after 4 weeks.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Tehsil Head Quarter Hospital Daska through consecutive sampling technique on 42 patients which will be allocated using computer generated sampling (random number table) into Group A and Group B. Group A will be treated with Postisometric relaxation technique and Group B will be treated with Static stretching technique. Postisometric relaxation will be performed with the frequency of 5 times, such that it includes (30 isometric contraction of the muscle to be stretched for 10 seconds, followed by rest period of 5 seconds and then a stretch of 10 seconds hold. Stretching exercise will be performed with 30 second hold and with 5 repetitions. All Exercises will be performed 3 times per week for total of 4 weeks. Outcome measures will be conducted through pain, range of motion, disability and muscle length after 4 weeks. Data will be analyzed during SPSS software version 25. The normality of data will be assessed by Shapiro-wilk test after which it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females.
* Age range of 24-59 years.
* Neck and medial border scapular pain for at least 3 months.
* NPRS score greater than 3.
* Reduced side flexion and rotation of neck.
* Symptoms persisted for at least 3 months.
* Positive levator scapulae length test.
* Have suffered from myofascial pain

Exclusion Criteria:

* Neuropathies.
* Vertebral fractures.
* Pregnancy.
* Fibromyalgia.
* Cancer.
* Traumatic neck injury.
* Previous cognitive and functional disorders.
* Coagulopathy(

Ages: 24 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-01-24 (Estimated); Study Completion 2025-02-24 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Pre & Post 6 weeks
  Numeric Pain Rating Scale
Disability Level | Pre & Post 6 weeks
  Neck Disability Index
Range of Motion | Pre & Post 6 weeks
  Goniometer
Muscle Length | Pre & Post 6 weeks
  Levator Scapulae Index

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Tehsil Headquarter Hospital Daska, Daska Kalan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No